CLINICAL TRIAL: NCT04917848
Title: Tele-Geriatric Oncology Program: Geriatric Assessment Via Telemedicine for Older Adults With Cancer
Brief Title: A Study of a Telemedicine Program for Older Adults With Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-200
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Cancer
Keywords: Geriatric Oncology Program; Geriatric Assessment; Telemedicine; Tele-Geriatric Oncology Program; 21-200; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Older adults with cancer (Experimental): Participants will be 70 years old or older with a diagnosis of gastrointestinal or gynecological cancer. Participants will be receiving or about to receive medical cancer treatment (e.g., chemotherapy, immunotherapy, targeted therapy, biological agents)
  Interventions: Other: Tele-Geriatric Oncology program

INTERVENTIONS:
Other: Tele-Geriatric Oncology program — Participants will be scheduled to meet with a Geriatric Nurse Practitioner (GNP) or Geriatric Registered Nurse (GRN) via the program's telemedicine platform. The telemedicine encounters with the GNP/GRN may occur every 2 weeks over 3 months, for a total of 6 visits. Visits 1 and 6 are mandatory, and visits 2-5 are on an as needed basis.

SUMMARY:
The purpose of this study is to find out if a telemedicine program for older adults in cancer treatment is a practical way to understand and meet these participants' unique needs. Telemedicine is the use of secure video technology on a desktop computer, laptop, smartphone, or tablet to provide and receive healthcare from a distance. The telemedicine program used in this study is called a tele-geriatric oncology program. It involves the participant and a study nurse meeting by videoconferencing during 2-6 telemedicine visits. As part of the program, the participant and the study nurse will discuss the participant's symptoms and aging-related needs.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 or older
* Gastrointestinal or gynecological cancer.
* Receiving or about to receive medical cancer treatment (e.g., chemotherapy, immunotherapy, targeted therapy, biological agents)

Exclusion Criteria:

* Inability of the patient or caregiver to read or comprehend English
* No internet connection at home
* No electronic device with videoconferencing capability

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Tele-Geriatric Oncology Program | 18 months
  We will report the proportion (and CI) of optional telemedicine visits attended by enrolled participants out of the total number of scheduled optional telemedicine encounters. As participants could have multiple scheduled optional appointments and these appointments for the same participant would be correlated, the confidence interval will be calculated based on bootstrapping our original sample.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Korc-Grodzicki, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org